CLINICAL TRIAL: NCT01567332
Title: Evaluation of Walking After Repetitive Transcranial Magnetic Stimulation (rTMS) Inhibitory 1Hz in Vascular Hemiplegia.
Acronym: rTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: BRD/10/04-P
Record Dates: First submitted 2012-03-26; First posted 2012-03-30 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rTMS active (Experimental)
  Interventions: Device: SHAM - MagproR30 - DGM-512 - 9016E0741 - Tonika elektronics A/S - Active coil
- rTMS inactive (sham) (Placebo Comparator)
  Interventions: Device: SHAM inactive - MagproR30 - DGM-512 - 9016E0741 - Tonika elektronics A/S - Inactive coil

INTERVENTIONS:
Device: SHAM - MagproR30 - DGM-512 - 9016E0741 - Tonika elektronics A/S - Active coil — For each patient, stimulation inactive (sham) and 1 Hz stimulation activates the healthy motor cortex (randomization). Active or sham session: Each session includes a series of 5 sessions of 20 'weekly (daily for 5 d) evaluation and pre-rTMS (T0 within 6 h before the procedure) and 1h post-rTMS (T1), at J8 (T2) and J21 (T3).
  6-week interval between two sessions.
  Arms: rTMS active
Device: SHAM inactive - MagproR30 - DGM-512 - 9016E0741 - Tonika elektronics A/S - Inactive coil — For each patient, stimulation inactive (sham) and 1 Hz stimulation activates the healthy motor cortex (randomization). Active or sham session: Each session includes a series of 5 sessions of 20 'weekly (daily for 5 d) evaluation and pre-rTMS (T0 within 6 h before the procedure) and 1h post-rTMS (T1), at J8 (T2) and J21 (T3).
  6-week interval between two sessions.
  Arms: rTMS inactive (sham)

SUMMARY:
Recovery of neurological deficits after stroke results from a reorganization of cortical activities, possibly through brain plasticity. Repetitive Transcranial Magnetic Stimulation (rTMS-MagproR30) produces changes in cortical excitability, generates phenomena of neuroplasticity. Its use to improve function after stroke, particularly of the upper limb, was validated. The investigators propose to evaluate in a prospective pilot against placebo, the benefit of rTMS at low frequency (1Hz) on the unaffected hemisphere in the short and medium term, especially on walking function and spasticity in patients with sequelae of cerebral infarction in the MCA territory with gait disturbance and motor weakness of the upper limb.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years of two sexes
* Cerebral infarction older than 12 months
* NIH score > 4
* Patient able to walk with or without technical assistance, Rankin score greater than or equal to 3
* No changes can interfere with treatment of spasticity in the 3 months preceding the study (benzodiazepines, baclofen, dantrolene, botulinum toxin ...)
* No history of generalized epilepsy unbalanced
* Free and informed consent signed by the patient
* MRI with ancient anatomical sequence confirming the accident sylvian

Exclusion Criteria:

* Stroke with motor sequelae of cerebral infarction prior to qualifying
* Alteration of the course prior to stroke
* Generalized epilepsy unbalanced
* Arrhythmias untreated
* Injection of botulinum toxin in the previous 4 months of randomization and 2 months after randomization
* Severe aphasia or cognitive impairment that interferes with the understanding of the tasks
* Presence of ferromagnetic material intracranial
* Pacemaker

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Spontaneous walking speed of 10 meters. The evaluation of the primary endpoint is blind to the stimulation | 3 months
  Spontaneous walking speed (comfortable) to 10 meters. The gain on the walking speed of 10 meters will be appreciated by an independent evaluator, blinded to randomization.
  The evaluation will be made on day 1 pre (T0) and post-stimulation (T1) (for 6 hours before and after 1 h), at D8 (T2) and J21 (T3) for 2 sessions (sham and active) .

SECONDARY OUTCOMES:
Distance covered in 6 min | 3 months
- Study of the march by AQM (Gait Deviation Index) | 3 months
  Measurement parameters spatiotemporal, kinematic and kinetic walking on day 1 pre-test, J8, J21 of the two phases.
  This measurement is performed using 4 cameras and markers installed in the room where runs quantified analysis of the march.
  Patients are fitted with reflective markers so that their movements are recorded and then digitized
- Consequence of lower limb spasticity (Modified Ashworth Scale of the quadriceps and triceps surae) | 3 months
  Used to describe a subjective rate of increase in resistance or tone perceived by an examiner when a member engages in the mobility sector. Coast of the score 0-4 (0 no strength, no mobility possible, 4). The scale is used to measure the first tone. Its reproducibility is quite low but it is the scale used and accepted. It is brief and feasible (no equipment, but requires training).Will be measured pre and post test J1, J8 and J21 of the two phases.
Analytical and functional recovery of the lower limb (Fugl-Meyer Scale, the FIM score) | 3 months
  The scale sensorimotor Fugl-Meyer: widely used in the literature, gold standard. The evolution motor is well defined. First part to obtain three subscores: MS (33 items, side 0 to 66), MI (17 items sides from 0 to 34), equilibrium (7 items sides from 0 to 14). The score can be used in total or subgroup. It requires 30 to 45 minutes with a trained evaluator. It can easily be used in clinical practice. A change in score <10 may be due to simple measurement error and may not reflect a significant change in motor skills.
  Will be measured pre and post test J1, J8 and J21 of the two phases.
Analytical and functional recovery of upper limb (Fugl-Meyer score and French arm test) | 3 months
  The Frenchay Arm Test: This test, rapid (5 min) includes five tasks rated 0 or 1, requiring the use of one or both hands: draw a line, then install a lift cylinder, lift and then rest a glass of water, remove and replace a clothespin and combing. The score ranges from 0 to 5. The FAT is used to evaluate both the proximal motor skills, manual dexterity and bimanual coordination. It is validated in hemiplegic, reproduced over time and between observers, but its ceiling and floor effects are very important. Will be measured pre and post test J1, J8 and J21 of the two phases.
Patient satisfaction and quality of life on a visual analog scale and the SF 36. | 3 months
  Is a generic health scale created to measure health status in the general population. It includes 36 items organized into eight dimensions, physical functioning, physical limitations, pain, social functioning, mental health, emotion, vitality, general health perceptions. It includes two questions to estimate the change of health status on the past four weeks. The test is validated, it is a simple questionnaire and short of 10 minutes (acceptability).It requires no training to administer. It can be done by mail (Feasibility).She will be provided on D8 of the two phases.

CONTACTS AND LOCATIONS:
Overall Officials: Angélique STEFAN, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Dr Angelique STEFAN, Nantes, France